CLINICAL TRIAL: NCT05473663
Title: A 6-month, Double-blinded, Sham-controlled Clinical Trial Assessing the Clinical Usefulness of Radiofrequency Ablation for Chronic Knee Pain After Total Knee Arthroplasty
Brief Title: Radiofrequency Ablation After Total Knee Arthroplasty
Acronym: RACKTKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Boston University (Other); Tufts Medical Center (Other); Rheumatology Research Foundation (Other)
Responsible Party: Principal Investigator, Timothy McAlindon, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00001815
Record Dates: First submitted 2022-07-18; First posted 2022-07-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Knee Pain
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Radiofrequency Ablation (Active Comparator): Patient undergoing genicular nerve radiofrequency ablation.
  Interventions: Device: Radiofrequency Ablation
- Sham (Sham Comparator): Patient undergoing sham.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Radiofrequency Ablation — Genicular nerve RFA is a standard outpatient procedure using fluoroscopic guidance to ensure accurate placement of the radiofrequency cannula. After placement of the radiofrequency cannula, nerve stimulation is performed to confirm proper position and ensure that the cannula is not too close to motor fibers. One mL of 2% lidocaine is placed at each of the cannulas. The RFA treatment is then proceeded by rhizotomizing each genicular nerve at 80°C for 90 seconds with a 15-second ramp-up.
  Arms: Radiofrequency Ablation
Device: Sham — Is performed identically to the active treatment but without the application of the RFA current
  Arms: Sham

SUMMARY:
The purpose of this study is to assess how clinically useful and safe genicular nerve radiofrequency ablation is in people with chronic pain after total knee arthroplasty performed for osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible individuals over 18 years of age in general good health apart from their chronic knee pain
2. At least one year post-TKA
3. Report of chronic knee pain classified using a standard question about the presence of "pain, aching, or stiffness in the knee on most days for at least one month during the prior 6 months"
4. In an unacceptable symptom state classified using a validated question: "Think about all consequences of your arthroplasty in the last week. If you were to remain for the rest of your life as you were during the last week, would the current state be acceptable or unacceptable for you?"
5. Willingness to complete all the study procedures, including a daily pain NRS, AE, and medication usage questions via daily notification
6. Subjects must have read and understood the informed consent form (ICF), and must have signed and dated it prior to any study-related procedure being performed

Exclusion Criteria:

1. Pregnant women, breastfeeding women, and women who are not post-menopausal (defined at 12 months with no menses without an alternative medical cause) or permanently surgically sterile (includes hysterectomy, bilateral salpingectomy, and bilateral oophorectomy)
2. Women who are not post-menopausal or permanently surgically sterile who are sexually active, and who are not willing to use birth control as outlined in Section 5.3.1 during the study period
3. Significant evidence of infection within the knee or radiographic evidence of prosthesis loosening as defined by the orthopedic surgeon
4. Individuals with pain exclusively located in the posterior knee, evaluated systematically using a validated Knee Pain Map
5. Individuals who do not achieve a 70% pain reduction following the initial prognostic block, consistent with clinical practice
6. Participation in a clinical research trial that included the receipt of an investigational product (IP) or any experimental therapeutic procedure within 30 days prior to the Screening Visit, or planned participation in any such trial
7. Use of anticoagulants and inability to withhold for three days prior to the study RFA procedure with clearance by the prescribing physician
8. Other conditions that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability by actively treated participants Outcome | 3 months
  Our a priori decision rule for acceptability of RFA will be that 50% of the actively treated participants respond affirmatively at the 3-month visit: "Would you recommend the treatment used in this study to someone in a similar situation with knee pain after a knee replacement?"
Safety Outcome | 6 months
  <2 serious adverse events among 20 actively treated participants. After enrollment, participants will complete training regarding the daily notification for daily adverse event monitoring. During the study, participants will be automatically prompted daily to report adverse events on their mobile device or home computer. If a participant does not complete adverse event monitoring daily, a member of the study team will contact them to troubleshoot.
  Additionally, a more thorough examination of patient safety will be conducted during the clinical exam in the 1-, 3-, and 6-month follow-up visits. Prosthesis safety will be assessed with skyline, lateral, and anteroposterior radiographs (e.g. aseptic loosening, osteolysis) at baseline and 6 months69. Serious adverse events will be consistent with our institution's IRB definitions and with a definition of serious adverse drug experience in FDA 21 CFR 312.32(a).
Efficacy Outcome | 3 months
  <5 number needed to treat to achieve a patient-acceptable symptom state. Patient acceptable symptom state will be defined with the following question: "Think about all consequences of your arthroplasty in the last week. If you were to remain for the rest of your life as you were last week, would the current state be acceptable or unacceptable for you?"61 Primary efficacy measure will be whether a participant considers themselves in an acceptable symptom state at the 3-month visit after the intervention. A <5 number is needed to treat to achieve a patient-acceptable symptom state.

SECONDARY OUTCOMES:
Pain Number Rating Score (NRS) | 6 months
  Change from baseline in daily pain number rating scale (NRS) scores via text or online platform until study completion. Min= 0, Max=10. Larger change in scores mean a better outcome.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 1-, 3-, and 6-month visits
  Change from baseline in the Knee Injury and Osteoarthritis Outcome Score (KOOS) Activities of Daily Living subscales at 1-, 3-, and 6-month visits. Questions measured from 0-4. Min = 0 (none), Max= 4 (extreme). Larger change in scores mean a better outcome.
Physical Activity Scale for the Elderly (PASE) | 1-, 3-, and 6-month visits
  Change from baseline in the Physical Activity Scale for the Elderly (PASE) at 1-, 3-, and 6-month visits. Measured based on frequency 0 (never)- 3 (often). Larger change in score means better outcome.
Quality of Life Measured using Knee Injury and Osteoarthritis Outcome Score Quality of Life (KOOS QOL) | 1-, 3-, and 6-month visits
  Change from baseline in the KOOS Quality of Life subscale at 1-, 3-, and 6-month visits. not at all- extreme. Larger change in score means better outcome.
Quality of Life Measured using Patient Reported Outcome Measurement Information System (PROMIS) Global 10 | 1-, 3-, and 6-month visits
  Change from baseline in the PROMIS Global 10 at 1-, 3-, and 6-month visits.
Walk Test | 1-, 3-, and 6-month visits
  Change from baseline in 20-meter walk test time at 1-, 3-, and 6 month visits
Chair Stand Test | 1-, 3-, and 6-month visits
  Change from baseline in chair stand speed at 1-, 3-, and 6- month visits
Daily Step Count | 1-, 3-, and 6-month visits
  Change from baseline in daily step count via Wearable Activity Monitor (i.e. Fitbit) averaged over the one week following 1-, 3-, and 6- month visits
Incidence of Pain Medication use | 1-, 3-, and 6-month visits
  Change from baseline in usage of pain medication for target knee pain at 1-, 3-, and 6- month visits. Measured using questionnaire.
Gait Analysis | 3 months
  An optional sub-study will assess change from baseline in spatiotemporal metrics of gait at the 3 month visit. . Data collected will include knee kinematics and kinetics using optical motion capture and spatiotemporal gait parameters using wearable inertial sensors. Larger change from baseline means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy E McAlindon, MD, MPH, Principal Investigator — UMass Worcester (UMass Chan Medical School)
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No